CLINICAL TRIAL: NCT01196481
Title: A Prospective,Open Labeled, Randomized Controlled Trial Comparing Carvedilol + VSL# 3 Versus Endoscopic Variceal Ligation for Primary Prophylaxis of Esophageal Variceal Bleeding in Cirrhotic Patients Non Responder to Carvedilol.
Brief Title: Carvedilol + VSL#3 Versus Endoscopic Variceal Ligation for Primary Prophylaxis of Esophageal Variceal Bleeding in Cirrhotic Patients Non Responder to Carvedilol.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ILBS PHT-04
Record Dates: First submitted 2010-09-04; First posted 2010-09-08 (Estimated); Last update posted 2020-05-15 (Actual); Status verified 2015-12

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carvedilol+VSL#3 (Experimental): Tablet Carvedilol 6.25 mg BD + VSL#3
  Interventions: Drug: Carvedilol+VSL#3
- Endoscopic Variceal Ligation (Active Comparator): Endoscopic Variceal Ligation every 3-4 weeks till variceal ligation
  Interventions: Drug: Carvedilol+VSL#3; Procedure: Endoscopic variceal ligation

INTERVENTIONS:
Drug: Carvedilol+VSL#3 — Tablet Carvedilol 6.25 mg BD & capsule VSL#3 1 TDS for 2 year
Procedure: Endoscopic variceal ligation — In the Endoscopic Variceal Ligation arm, Endoscopic Variceal Ligation will be performed using multibander devices by senior fully trained endoscopists or under their direct supervision. Varices will be banded starting at the gastroesophageal junction moving proximally upward in a spiral fashion. Patients will undergo Endoscopic Variceal Ligation every 3-4 weeks until eradication. Eradication is defined as the absence of varices or presence of grade I esophageal varices. Following eradication, the interval for the next endoscopy will be every 3 months to look for recurrence of varices. Endoscopic Variceal Ligation sessions would be repeated for the recurrent varices if they are sufficiently large.
  Arms: Endoscopic Variceal Ligation

SUMMARY:
Patients of cirrhosis will be enrolled who have large esophageal varices, which have never bled. After successful screening baseline hepatic venous pressure gradient (HVPG) will be measured. Tablet carvedilol 3.125 mg BD for 1 week will be started. It will be increased to 6.25 mg BD and continued for next 7 weeks. After completion of 8 weeks the hepatic venous pressure gradient (HVPG) will again be measured to find out responders (hepatic venous pressure gradient ≥20% reduction from baseline or absolute value of hepatic venous pressure gradient <12 mm Hg) and non responders (hepatic venous pressure gradient <20% reduction).The responders will be excluded from the study while the non responders will be randomize into carvedilol+VSL#3 versus Endoscopic Variceal Ligation.

ELIGIBILITY:
Inclusion Criteria:

* Patients of cirrhosis with portal hypertension aged 18 to 75 years who have large esophageal varices with or without red color signs and have not bled previously.

Exclusion Criteria:

* Any contra-indication to beta-blockers
* Coagulopathy with INR >1.8 at the time of enrollment
* Any Endoscopic Variceal Ligation or sclerotherapy within last 3 months
* Any past history of surgery for portal hypertension
* Significant cardio or pulmonary co-morbidity
* Any malignancy
* Refusal to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Development of first variceal bleeding | 1 Year

SECONDARY OUTCOMES:
Survival | 1 Year
Reduction in Portal pressure | 1 Year
Time to bleed | 1 Years
Adverse events | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Shiv Kumar Sarin, MBBS, MD, DM, Principal Investigator — Institute of Liver & Biliary Sciences (ILBS)
Locations (1):
- Institute of Liver & Biliary Sciences (ILBS), New Delhi, National Capital Territory of Delhi, India